CLINICAL TRIAL: NCT02282592
Title: Metabolic Syndrome and Female Breast Cancer: a Case-control Study in Southern Brazil
Brief Title: Metabolic Syndrome and Female Breast Cancer
Status: Completed | Type: Observational
Sponsor: Catholic University of Pelotas (Other)
Responsible Party: Principal Investigator, Rafaela Bulow Bergmann, Master in Health and Behavior, Catholic University of Pelotas
Other Study IDs: 481.165
Record Dates: First submitted 2014-10-17; First posted 2014-11-04 (Estimated); Last update posted 2014-11-04 (Estimated); Status verified 2014-10

CONDITIONS: Breast Cancer
Keywords: Metabolic syndrome; case-control study; Breast cancer
MeSH Terms: conditions — Breast Neoplasms; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- Cases: newly diagnosed (within 6 months) breast cancer patients, before adjuvant or neoadjuvant treatment.
  Interventions: Other: Observation about the presence of metabolic syndrome
- Controls: patients without any malignant disease, matched for age an menopausal status with cases.
  Interventions: Other: Observation about the presence of metabolic syndrome

INTERVENTIONS:
Other: Observation about the presence of metabolic syndrome

SUMMARY:
The role among metabolic syndrome and breast cancer risk is not well understood and must be further explored. The objective of this study is to evaluate the association between metabolic syndrome and breast cancer in Southern Brazil. In this case-control study, breast cancer patients and controls without malignant disease, matched for age (±5 years) and menopausal status, were interviewed and asked to make a glucose, HDL-cholesterol and triglycerides test. Waist circumference and blood pressure were measured using standardized procedures. Metabolic Syndrome was considered by NCEP ATP III (2001) and IDF (2006) definitions. Cases and controls were compared in relation to the presence of diagnosed MetS (yes/no), number of metabolic abnormalities identified (1 to 5) for each definition, and according to each metabolic abnormality cutoff point.

ELIGIBILITY:
Inclusion Criteria:

* For cases: having newly diagnosed breast cancer without adjuvant or neoadjuvant treatment;
* For controls: having no evidence of cancer; be matched for age and menopausal status with controls

Exclusion Criteria:

* Women with a recidivated tumor, HIV infection, renal, heart or liver disease, hypothyroidism or hyperthyroidism, mobility or neurological limitations, chronicle use of corticosteroids, pacemakers or identified with severe edema were excluded.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Between December 2013 and August 2014, newly diagnosed (within 6 months) BC female patients referred to the oncology sector of the Teaching Hospital of the Federal University of Pelotas and to the Radiotherapy and Oncology Center of Santa Casa de Misericordia of Pelotas were invited to the study, before starting any adjuvant or neoadjuvant treatment. Women with a recidivated tumor, HIV infection, renal, heart or liver disease, hypothyroidism or hyperthyroidism, mobility or neurological limitations, chronicle use of corticosteroids, pacemakers or identified with severe edema were excluded. For each cancer case, one female control should be matched for age (± 5 years) and menopausal status (pre and post-menopausal). Apart from being free from all the exclusion criteria used for BC cases, controls should also have no signs of malignant disease. These women were invited to participate in the study while frequenting the Gynecologic Ambulatory of the same institutions, in the same period.
Sampling Method: Non-Probability Sample
Enrollment: 164 (Actual)
Dates: Start 2013-11; Primary Completion 2014-08 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Odds Ratio for Breast Cancer according to the presence of Metabolic Syndrome and its components | Participants will be evaluated only once before the first appointment with the oncologist (cases with a biopsy) and gynecologist (controls). The blood test results for Metabolic Syndrome parameters were collected in an expected average of 30 days.